CLINICAL TRIAL: NCT06187558
Title: Suspension of the Pelvic and Abdominal Organs During Minimally Invasive Surgery
Status: Completed | Type: Observational
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Stefano Angioni, Professor, University of Cagliari
Other Study IDs: LPS SUSPENSION
Record Dates: First submitted 2023-10-25; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Endometriosis; Pelvic Prolapse; Endometrium Cancer
Keywords: Organ Suspension Techniques; Ovariopexy; Laparoscopic
MeSH Terms: conditions — Endometriosis; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pelvic Organ Suspension Patients: This group comprises patients who have undergone multiport or single-port access laparoscopic surgery (SPAL) at the Tertiary referral University Hospital of Cagliari, Italy. These patients suffer from benign (like endometriosis, pelvic prolapse) or malignant (like endometrial cancer) gynecological diseases. During their surgery, they have experienced at least one instance of the described pelvic organ suspension technique using an adjustable tension suture tied to a Foley catheter fragment for organ suspension.
  Interventions: Procedure: Pelvic and abdominal organ suspension technique

INTERVENTIONS:
Procedure: Pelvic and abdominal organ suspension technique — The intervention involves a unique organ suspension technique tailored for minimally invasive gynecologic surgeries. A fragment of a Foley catheter (2 cm of a 1 Fr/Ch) is tied at the end of an absorbable 2-0 Polyglactin suture with a straight needle to create the suspension device. This suture is introduced into the pelvic cavity via an ancillary port. It's designed to penetrate organs such as the ovary, posterior peritoneum, vesico-uterine peritoneum, or bowel. Once the suture is retrieved by passing it through the abdominal wall and pulled so that the Foley segment faces the organ's surface, it's secured using a Kelly clamp. This setup eliminates the need for a knot and offers the surgeon the flexibility to adjust the suspension tension as required.

SUMMARY:
The goal of this retrospective observational study is to evaluate the efficacy, safety, and practicality of an organ suspension technique with adjustable tension suture in facilitating minimally invasive gynecologic surgeries at the University Hospital of Cagliari, Italy. The main questions it aims to answer are:

* Is the organ suspension technique using adjustable tension suture both cost-effective and practical for minimally invasive gynecologic surgeries?
* How safe, effective, and feasible is this suspension technique when applied to patients with benign or malignant gynecological diseases undergoing laparoscopic surgery?

Participants in this study underwent laparoscopic surgery involving the organ suspension technique, which includes:

* The use of a modified Foley catheter and Polyglactin suture for organ suspension.
* The collection of preoperative and postoperative data, such as operation times, blood loss, hospital stay duration, and short-term postoperative complications.

This study does not include a comparison group, focusing instead on the direct outcomes and experiences of the participants who underwent the specified surgical technique.

DETAILED DESCRIPTION:
This retrospective observational study, conducted at the University Hospital of Cagliari in Italy, is focused on providing a comprehensive evaluation of an innovative organ suspension (OS) technique using an adjustable tension suture in minimally invasive gynecologic surgery. The primary aim of the study is to determine the safety, efficacy, and feasibility of this technique, especially in the context of both benign and malignant gynecological diseases.

The OS technique is characterized by its unique use of a 2 cm segment of a 1 Fr/Ch Foley catheter, which is tied at the end of an absorbable 2-0 Polyglactin suture equipped with a straight needle. This assembly is strategically inserted into the pelvic cavity through an ancillary port. The primary function is to suspend critical organs such as the ovary, posterior peritoneum, vesico-uterine peritoneum, or bowel, facilitating better surgical access and maneuverability. The suture, once in place, is retrieved and pulled through the abdominal wall, positioning the Foley catheter such that it faces the surface of the suspended organ. This setup is secured using a Kelly clamp without a knot, allowing the surgeon to adjust the tension of the suspension as required during the surgery.

The study's participants comprise patients who underwent laparoscopic surgery for various gynecological conditions, including benign issues like endometriosis and pelvic prolapse, as well as malignant diseases such as endometrial cancer. The data collection for these participants is twofold: preoperative and postoperative. Preoperatively, the study gathers information on age, clinical history, symptoms, the location of the pathology, operation times, and blood loss. Postoperatively, the focus shifts to the number of days of hospital stay and the incidence of short-term postoperative complications, defined as those occurring within 30 days of the surgery.

By thoroughly analyzing this data, the study aims to answer critical questions regarding the cost-effectiveness, practicality, safety, and effectiveness of the OS technique. This could potentially lead to significant advancements in the field of minimally invasive gynecologic surgery, offering insights into more effective and patient-friendly surgical approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent multiport or single-site-port laparoscopic surgery with at least one transient pelvic organ suspension.
* Surgeries performed between March 2019 and May 2021.
* Surgeries conducted in the specified tertiary referral hospital.
* Patients who provided written informed consent for the surgical procedure and for the use of their personal data in scientific research.
* Availability of medical records and videos of surgeries for data collection.
* Patients who underwent surgery for one of the following conditions:
* Deep infiltrating endometriosis (DIE)
* Endometrial Cancer
* Pelvic prolapse treated by laparoscopic surgical procedure
* Single-port access laparoscopy for benign gynecological diseases
* Surgeries performed by either senior surgeon (S.A.) or junior surgeon (M.N.D).

Exclusion Criteria:

* Surgeries conducted outside the timeframe of March 2019 to May 2021.
* Surgeries not involving multiport or single-site-port laparoscopic surgery with pelvic organ suspension.
* Patients who did not provide written informed consent.
* Absence of medical records or surgery videos for data collection.
* Surgeries not performed in the mentioned tertiary referral hospital.
* Surgeries not primarily conducted for the specified indications (i.e., DIE, oncological disease, pelvic prolapse).
* Surgeries not performed by the listed surgeons (S.A. or M.N.D).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprised female patients who attended the University Hospital of Cagliari, a tertiary referral hospital. They underwent either multiport or single-site-port laparoscopic surgeries. The study retrospectively observed a total of 330 patients who had their surgeries between March 2019 and May 2021. Patients underwent surgery due to:
  Deep infiltrating endometriosis (DIE) Oncological disease Pelvic prolapse treated by laparoscopic surgical procedure Single-port access laparoscopy for benign gynecological diseases (SPAL)
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Safety of the Organ Suspension (OS)Technique | during the procedure
  Incidence of OS-Related Complications: Measurement of the rate of organ-specific complications and injuries during the Organ Suspension (OS) technique.
Efficacy of the Organ Suspension (Os) Tecnique | During the procedure
  Time required to achieve transient organ suspension, with comparison across organ types, surgeon experience levels, and patient BMI categories. Unit of Measure: Minutes to achieve suspension.
Rate of Laparotomy Conversion During OS Technique | during the procedure
  This measure assesses the frequency of conversion from the Organ Suspension (OS) technique to open laparotomy during surgery. The focus is to quantify how often the intended OS procedure is converted to a traditional laparotomy, indicating challenges or complications with the OS technique. Unit of Measure: Percentage of surgeries converted to laparotomy (%)

SECONDARY OUTCOMES:
Average Total Blood Loss in OS Technique | during surgery
  Measurement of the average total blood loss during surgery using the OS technique. Unit of Measure: Milliliters (ml)
Postoperative Analgesic Requirement | immediately after surgery
  Postoperative analgesic drug management in patients undergoing OS technique. Unit of Measure: Analgesic dosage (mg) and frequency of administration
Mean Duration of Hospital Stay Post-OS Technique | immediately after surgery
  Evaluation of the mean duration of hospital stay post-surgery, with significant differences highlighted based on the indication for surgery. Unit of Measure: Days

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Angioni, Principal Investigator — University of Cagliari
Locations (1):
- Division of Gynecology and Obstetrics Department of Surgical Sciences, University of Cagliari, Cagliari, Italy, Monserrato, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angioni S. New insights on endometriosis. Minerva Ginecol. 2017 Oct;69(5):438-439. doi: 10.23736/S0026-4784.17.04089-8. Epub 2017 May 25. No abstract available. PMID 28545294
- [Background] Chaichian S, Saadat Mostafavi SR, Mehdizadehkashi A, Najmi Z, Tahermanesh K, Ahmadi Pishkuhi M, Jesmi F, Moazzami B. Hyaluronic acid gel application versus ovarian suspension for prevention of ovarian adhesions during laparoscopic surgery on endometrioma: a double-blind randomized clinical trial. BMC Womens Health. 2022 Feb 11;22(1):33. doi: 10.1186/s12905-022-01607-2. PMID 35148732
- [Background] Chatzipapas I, Kathopoulis N, Kypriotis K, Samartzis K, Siemou P, Protopapas A. A simple technique for suspension and stabilization of retrieval bag and adnexa by anchoring to the abdominal wall. Clin Case Rep. 2021 Nov 19;9(11):e05056. doi: 10.1002/ccr3.5056. eCollection 2021 Nov. PMID 34840798
- [Background] Thompson R, Cesta M, Pasic R. Improved Exposure in Minimally Invasive Excision of Endometriosis with Temporary Ovarian Suspension Using Carter-Thomason CloseSure System, a Novel Technique. J Minim Invasive Gynecol. 2021 Oct;28(10):1678. doi: 10.1016/j.jmig.2021.05.004. Epub 2021 May 17. PMID 34015526
- [Background] Abuzeid OM, Hebert J, Ashraf M, Mitwally M, Diamond MP, Abuzeid MI. Safety and efficacy of two techniques of temporary ovarian suspension to the anterior abdominal wall after operative laparoscopy. Facts Views Vis Obgyn. 2018 Jun;10(2):71-79. PMID 31110645